CLINICAL TRIAL: NCT06335498
Title: A Further Study of the Clinical Performance of AFGen1
Brief Title: Further Study of AFGen1 Clinical Performance
Acronym: CS3
Status: Completed | Type: Observational
Sponsor: TriVirum, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 130-0008P
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Atrial Fibrillation; Afib; ECG
Keywords: ECG signal quality
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Wear AFGen1 for at least 7 days: Wear AFGen1 for 7 to 10 days. ECG co-measurement with 12 lead device at start and periodic measurements of ECG with AFGen1 during wear period
  Interventions: Device: ECG co-measurement; Device: Periodic ECG triggered measurement
- Misplacement Study Group: Wear AFGen1 device in misplaced position compared to wearing device in standard position as directed by instructions for use
  Interventions: Device: ECG co-measurement

INTERVENTIONS:
Device: ECG co-measurement — Measure ECG with 12 lead device at same time that AFGen1 is monitoring ECG
Device: Periodic ECG triggered measurement — Subject triggers AFGen1 to perform an extended measurement during wear period
  Groups: Wear AFGen1 for at least 7 days

SUMMARY:
AFGen1 is indicated for use on symptomatic or asymptomatic adults who are at risk of developing or who have atrial fibrillation, where a software assisted analysis of ambulatory ECG is needed to identify episodes of Afib. The purpose of this study is to establish further evidence for the clinical performance of AFGen1 on human participants.

DETAILED DESCRIPTION:
The primary purpose of this study is to demonstrate the ECG signal acquired by the AFGen1 device is of adequate quality and is suitable to support its intended use for the detection of Afib. This will be evaluated by comparing the ECG data acquired by AFGen1 to that acquired by an FDA cleared 12-lead ECG device using a Bland-Altman analysis of the R-R intervals and R amplitude measurements and Eigenvector magnitudes derived from principal component analyses of simultaneously captured waveforms measured by both devices by both devices. The ECG waveforms from both devices will also be adjudicated by 2 independent cardiologists. The study will also seek to demonstrate that there is no degradation in the quality of the ECG signal it acquires when the device is placed in an anticipated misplacement position to that directed by the instructions for use of the device. Finally the study will seek to confirm the adhesive performance of the device is appropriate to support its intended use per the requirements of sections 4.4 and 5.4 of ANSI AAMI EC12-1 . Another purpose of the study is to collect extended 5 minute ECG recordings by the subject periodically triggering the device while wearing the device for 7 (+3) days. This data will be used for product development purposes.

ELIGIBILITY:
Inclusion Criteria:

1. 18+ willing to sign the consent form

Exclusion Criteria:

1. Implanted pacemakers
2. Implanted cardioverter defibrillators
3. Implanted cardiac resynchronization devices
4. Potential life-threatening arrythmias
5. Physical or mental health conditions that would prevent the person from being able to follow instructions regarding participation in the study
6. Open wounds, abraded or irritated skin at the application site
7. Planned to undergo a MRI during the course of the study duration
8. Known or suspected to be pregnant
9. Student or employee of TriVirum

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study shall involve up to twenty (20) participants divided into 2 cohorts. The first study cohort will comprise up to fifteen (15) participants (at least 5 male and 5 female) who will wear the device for 7 days. The second cohort of five (5) participants will participate in the misplacement part of the study
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Bland-Altman Comparison | 1 day
  The waveform characteristics for both the 7- day wear and misplacement elements of this study, the limits of agreement (LoA) from the Bland-Altman analyses shall not exceed the the maximum allowed clinically significant difference between methods i.e. 80ms for R-R. 0.2 mV for R-peak amplitude) for 95% of the subjects on a per-subject basis.
Qualitative Evaluation | 1 day
  For the qualitative equivalence evaluation according to the two cardiologists confirmation of equivalence must be greater than 95%.
Adhesive performance | 7 to 10 days
  The overall average wear time for the device must be greater than 7-days.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Willis, BSN RN, Principal Investigator — Unafilliated
Locations (1):
- 1808 49Th St Ct NW, Gig Harbor, Washington, United States

IPD SHARING:
Plan to Share IPD: No